CLINICAL TRIAL: NCT02832219
Title: Medium-term Effects of Molecular Hydrogen on Metabolic Fitness in Obesity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Center for Health Sciences, Serbia (Other)
Responsible Party: Principal Investigator, Assoc. Prof. Sergej M. Ostojic, MD, PhD, Principal Investigator, Center for Health Sciences, Serbia
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: 16-AD
Record Dates: First submitted 2016-07-05; First posted 2016-07-14 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Obesity
Keywords: Overweight; Molecular hydrogen; Insulin
MeSH Terms: conditions — Obesity; Overweight; Insulin Resistance | interventions — Hydrogen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Molecular hydrogen (Experimental): Molecular hydrogen, tablet, 2 g/day, 4 weeks
  Interventions: Dietary Supplement: Molecular hydrogen
- Placebo (Placebo Comparator): Cellulose, tablet, 2 g/day, 4 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Molecular hydrogen
  Arms: Molecular hydrogen
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Molecular hydrogen (H2) effectively tackles obesity-related disorders in animal models yet no studies so far investigated the effectiveness of H2 for improving biomarkers of obesity in humans. In this double blind, placebo-controlled, crossover pilot trial, the investigators will evaluate the effects of H2 intervention on body composition, hormonal status, and mitochondrial function in middle age overweight women, with hydrogen administered orally for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* age > 55 years
* body mass index > 25 kg/m2

Exclusion Criteria:

* no history of H2 supplementation within the 4 weeks before study commenced
* no major chronic diseases, as evaluated by pre-participation health screening and clinical chemistry

Min Age: 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-01; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Body fat percentage change | Baseline vs. four weeks
  Baseline vs. four weeks

SECONDARY OUTCOMES:
Serum insulin change in IU/mL | Baseline vs. four weeks
  Baseline vs. four weeks

OTHER OUTCOMES:
Serum ghrelin change in IU/mL | Baseline vs. four weeks
  Baseline vs. four weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Health, Exercise and Sport Sciences, Belgrade, Serbia, Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ostojic SM. Molecular hydrogen: An inert gas turns clinically effective. Ann Med. 2015 Jun;47(4):301-4. doi: 10.3109/07853890.2015.1034765. Epub 2015 May 4. PMID 25936365
- [Background] Huang CS, Kawamura T, Toyoda Y, Nakao A. Recent advances in hydrogen research as a therapeutic medical gas. Free Radic Res. 2010 Sep;44(9):971-82. doi: 10.3109/10715762.2010.500328. PMID 20815764
- [Derived] Korovljev D, Trivic T, Drid P, Ostojic SM. Molecular hydrogen affects body composition, metabolic profiles, and mitochondrial function in middle-aged overweight women. Ir J Med Sci. 2018 Feb;187(1):85-89. doi: 10.1007/s11845-017-1638-4. Epub 2017 May 30. PMID 28560519